CLINICAL TRIAL: NCT02904577
Title: Indolent Non Follicular Lymphomas Prognostic Project - Prospective Collection of Data of Possible Prognostic Relevance in Patients With Indolent Non-follicular B-CELL Lymphomas
Brief Title: Indolent Non Follicular Lymphomas Prognostic Project
Status: Completed | Type: Observational
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Responsible Party: Sponsor
Other Study IDs: NF2010
Record Dates: First submitted 2016-09-06; First posted 2016-09-19 (Estimated); Last update posted 2025-08-08 (Actual); Status verified 2024-12

CONDITIONS: Indolent B-Cell Lymphomas
Keywords: Indolent B-Cell Lymphomas; prospective collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Central pathological review. The reviewed material will refer to both onset and eventual relapse.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Training and validation cohort: One cohort: from this cohort 2/3 of patients will be randomly separated after registration in training sample, to develop a prognostic model, and 1/3 in test sample, to validate the prognostic score obtained from the prognostic model.
  The training cohort aims to develop a prognostic model and a resulting score, on the basis of clinical, biochemical and blood count parameters, in patients with non-follicular indolent lymphomas.
  Intervention: any treatment, watch and wait policy included
  The validation cohort is aims to assess the prognostic score on a collected set of data in parallel but independently of the "sample training".
  Intervention: any treatment, watch and wait policy included
  Interventions: Other: Any treatment, watch and wait policy included

INTERVENTIONS:
Other: Any treatment, watch and wait policy included — Patients registered in the study despite their planned treatment, watch and wait policy included. The "planned treatment" mentioned in the protocol is just the ideal approach proposed by investigators.The treatment can change depending on the evolution of the disease, without this affects the study's purposes.

SUMMARY:
Prospective collection of data of possible prognostic relevance in patients with indolent non - follicular B-CELL Lymphomas.

DETAILED DESCRIPTION:
The present study is designed as a prospective collection of information potentially useful to predict the prognosis of newly diagnosed patients with non-follicular low grade B-cell lymphoma.

The study is aimed to verify whether a prognostic collection of data would allow the development of a more accurate prognostic assessment for non-follicular low grade B-cell lymphomas.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed diagnosis of non-follicular low grade B-cell lymphoma

   * Splenic MZL (bone marrow histology and/or spleen tissue)
   * Extranodal MZL of MALT (tissue biopsy)
   * Nodal MZL (lymph node biopsy)
   * Lymphocytic lymphoma (lymph node biopsy)
   * Lymphoplasmacytic lymphoma (bone marrow histology or lymph node biopsy)
   * CD5-negative low grade B-cell lymphoma (bone marrow histology)
2. Age over 18
3. Written informed consent

Exclusion Criteria:

1. None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histologically confirmed diagnosis of non-follicular low grade B-cell lymphoma.
Sampling Method: Non-Probability Sample
Enrollment: 370 (Estimated)
Dates: Start 2011-09 (Actual); Primary Completion 2024-12 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Progression-free survival for the treated cohort | September 2024 (13 years)
  Progression free survival (PFS) will be measured from the date of randomization to the date of documented first occurrence of disease progression or relapse or to the date of death from any cause. Patients who are lost to follow up will be censored at their last assessment date.

SECONDARY OUTCOMES:
Progression-free survival for the untreated cohort | September 2024 (13 years)
  Progression free survival (PFS) will be measured from the date of randomization to the date of documented first occurrence of disease progression or relapse or to the date of death from any cause. Patients who are lost to follow up will be censored at their last assessment date.
Overall survival | September 2024 (13 years)
  Overall survival (OS) is defined as the time from the study entry until the date of death irrespective of cause. Patients who have not died at the time of end of the whole study , and patients who are lost to follow up , will be censored at the date of the last contact.
Event-free survival | September 2024 (13 years)
  Event Free Survival (EFS) is measured from the time from study entry to any treatment failure including disease progression, or discontinuation of treatment for any reason (eg, disease progression, toxicity, patient preference, initiation of new treatment without documented progression) or death from any cause.
Remission rate with initial therapy | September 2017 (Six years)
  Remission rate (RR) is defined as the number of complete and partial remission (CR and PR) after the completion of the first line of treatment.
Epidemiology | September 2016 (Five years)
  Will be collected the risk factors potentially associated to the outcome of indolent non follicular lymphomas (clinical status, biochemistry, hemochrome, HCV, HBV and autoimmnity markers). Will be collected the risk factors potentially associated to the outcome of indolent non follicular lymphoma (clinical status, biochemistry, hemochrome, HCV, HBV and autoimmunity markers). Those risk factors will be utilized to obtain a prognostic model (prognostic index) from the Cox proportional hazard regression and, finally, a prognostic score grouping the prognostic index in at least three group of risk (low, intermediate, high risk).
Time dependent analysis for patients in Watch & Wait policy. | September 2024 (13 years)
  In WW group the start of treatment will be treated as a time-varying covariate in Cox proportional hazard regression.
Remission rates with second and subsequent lines of therapy | September 2024 (13 years)
  Remission rate (RR) is defined as the number of CR and PR after the second and subsequent lines of therapy, due to progression disease.

CONTACTS AND LOCATIONS:
Overall Officials: Arcaini Luca, MD, Study Chair — Divisione di Ematologia IRCCS Policlinico S. Matteo Pavia
Locations (46):
- Vienna Univ Med Int I, Vienna, Austria
- Brazil (3):
  - Center of Hematology and Hemotherapy, UNICAMP, University of Campinas, Campinas
  - Universidade Federal Do Rio de Janeiro, Rio de Janeiro
  - São Paulo-Santa Casa Medical School, São Paulo
- Hospital Saint-Louis, Paris, France
- Italy (39):
  - UO Oncoematologia Ospedale Umberto I, Pagani, Salerno
  - Oncologia Medica A - Centro di Riferimento Oncologico, Aviano (PN)
  - UO Ematologia con Trapianto Policlinico Consorziale, Bari
  - USC Ematologia Ospedali Riuniti di Bergamo, Bergamo
  - Ematologia e CTMO Ospedale Businco, Cagliari
  - UOC Ematologia, Azienda Ospedaliera Garibaldi P.O. Nesima, Catania
  - US Oncoematologia- Ospedale Valduce, Como
  - Unità Operativa Complessa di Ematologia - AO di Cosenza, Cosenza
  - UO Ematologia, PO Vito Fazzi, Lecce
  - Ematologia Ospedale Madonna delle Grazie, Matera
  - SC. Ematologia. Osp. Riuniti Papardo Piemonte, Messina
  - Dipartimento di Oncoematologia Ospedale San Raffaele, Milan
  - SC Ematologia AO Niguarda Ca' Granda, Milan
  - UO Ematologia, AO San Carlo Borromeo, Milan
  - UO Oncologia Medica, Ospedale San Paolo, Milan
  - UOC Ematologia 1/CTMO, Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan
  - Dipartimento di Oncologia ed Ematologia Università di Modena e Reggio Emilia, Modena
  - Clinica Ematologica AO San Gerardo di Monza, Monza
  - SCDU Ematologia - AOU Ospedale Maggiore, Novara
  - Istituto Oncologico Veneto IRCCS, Padua
  - Ematologia e CTMO Ospedale Maggiore di Parma, Parma
  - Ematologia IRCCS Policlinico S. Matteo di Pavia, Pavia
  - Dipartimento di Ematologia Ospedale Civile Spirito Santo Pescara, Pescara
  - UO Ematologia AOU S. Chiara Pisa, Pisa
  - Divisione di Ematologia - Azienda Ospedaliera Bianchi Melacrino Morelli, Reggio Calabria
  - SC Ematologia Arcispedale Santa Maria Nuova, Reggio Emilia
  - UO Ematologia e Trapianto Cellule Staminali, IRCCS, Centro di riferimento Oncologico di Basilicata, Rionero in Vulture
  - Ematologia Università Campus Biomedico, Roma
  - Ematologia Università Roma La Sapienza, Roma
  - UOSD DH Ematologia Ospedale San Eugenio, Roma
  - Dipartimento di Oncologia Medica ed Ematologia Istituto Humanitas, Rozzano (MI)
  - UOC Medicina Interna MO DH Oncologico, Sassuolo
  - UOC Ematologia, AOU Senese, Siena
  - Ematologia PO SG Moscati, Taranto
  - SC Oncoematologia con autotrapianto AO S. Maria Terni, Terni
  - SC Ematologia Universitaria, AO Città della Salute e della Scienza, Torino
  - SC Ematologia, AO Città della Salute e della Scienza, Torino
  - Unità operativa Complessa Ematologia - Azienda Ospedaliera Ospedale di Circolo e Fondazione Macchi, Varese
  - Divisione di Ematologia, Ospedale San Bortolo, Vicenza
- LISBOA-IPO "Francisco Gentil", Lisbon, Portugal
- National Cancer Institute of Health Ukraine, Kiev, Ukraine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Luminari S, Merli M, Rattotti S, Tarantino V, Marcheselli L, Cavallo F, Varettoni M, Bianchi B, Merli F, Tedeschi A, Cabras G, Re F, Visco C, Torresan Delamain M, Cencini E, Spina M, Ferrero S, Ferrari A, Deodato M, Mannina D, Annibali O, Rago A, Orsucci L, Defrancesco I, Frigeni M, Cesaretti M, Arcaini L. Early progression as a predictor of survival in marginal zone lymphomas: an analysis from the FIL-NF10 study. Blood. 2019 Sep 5;134(10):798-801. doi: 10.1182/blood.2019001088. Epub 2019 Jul 10. PMID 31292118